CLINICAL TRIAL: NCT07250282
Title: Impact of Virtual Reality on Patients' Anxiety and Pain During Implantation of Cardiac Pacemakers, Implantable Cardioverter-defibrillators, or Cardiac Resynchronization Therapy: a Randomized Controlled Study
Brief Title: Impact of Virtual Reality on Anxiety and Pain During Implantation of Cardiac Implantable Electronic Devices (CIED)
Acronym: CIED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammed Kurt (Other)
Responsible Party: Sponsor-Investigator, Muhammed Kurt, Attending physician, Department of Cardiology and Vascular Medicine, University Hospital Essen, University Hospital, Essen
Organization: University Hospital, Essen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-11442-BO
Record Dates: First submitted 2025-11-17; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Anxiety; Pain
Keywords: CIED; Pacemaker; Virtual reality; ICD; CRT
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The patients in control arm received the standard preoperative care using local anesthesia
- intervention group (Experimental): The patients in intervention arm received a virtual reality headset in addition to the standard care using local anesthesia
  Interventions: Other: Virtual reality headset

INTERVENTIONS:
Other: Virtual reality headset — A virtual reality headset was used during the study with the purpose of distracting the patients from painful and stressful stimuli in the operation room to decrease their anxiety and pain perception
  Arms: intervention group

SUMMARY:
Purpose:

This study aimed to evaluate whether virtual reality technology positively affects patients' pain and anxiety throughout the entire procedure of implantation of cardiac pacemakers, defibrillators, or cardiac resynchronisation therapy.

DETAILED DESCRIPTION:
Methods:

From January 2024 to Mai 2025, 100 Patients undergoing implantation of cardiac single-chamber or dual-chamber pacemakers or defibrillators and cardiac resynchronisation therapy were included in this study. Patients were randomly assigned to either a control group (n=50) or an intervention group (n=50). The control group received standard preoperative care and local anaesthesia using lidocaine. A virtual reality headset was used in the intervention group in addition to the standard preoperative care and local anaesthesia during the procedure. The procedure was performed in all patients using standard preparation and cephalic vein cutdown. The State-Trait Anxiety Inventory-State (STAI-S) questionnaire was filled out by patients pre- and postoperatively to determine their anxiety levels before and during the procedure.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18 years
* Indication for implantation of a cardiac pacemaker, ICD, or CRT device due to one of the following:
* Complete heart block (AV block III°)
* Symptomatic bradycardia due to sinus node dysfunction
* Tachy-brady syndrome
* Atrial fibrillation with slow ventricular rate
* Symptomatic bradycardia due to AV block II° type Mobitz
* Secondary prevention of sudden cardiac death due to ventricular tachycardia
* Primary prevention in patients with heart failure with reduced ejection fraction
* Primary prevention in patients with heart failure with reduced ejection fraction and complete left bundle branch block
* "Pace and ablate" strategy for therapy-resistant persistent atrial fibrillation
* Need to Upgrade to CRT-P due to a high percentage of right ventricular pacing

Exclusion Criteria:

* Intolerance or inability to wear the VR headset
* Significant language barrier preventing consent or cooperation
* Need for deep sedation or general anesthesia for the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Baseline to perioperative anxiety change using State-Trait Anxiety Inventory-State (STAI-S) questionnaire score pre- and periprocedurally (Score range between 20 - 80, higher score means greater state anxiety) | From enrolment to the first postoperative day
  The anxiety reduction of patients from preprocedural to periprocedural state defined as reduction in STAI-S Scores pre and periprocedural was compared between the groups as the primary endpoint of the study

CONTACTS AND LOCATIONS:
Locations (1):
- West german heart and vascular center, University hospital Essen,, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided